CLINICAL TRIAL: NCT00904644
Title: Raltegravir Use in the Swiss HIV Cohort Study (SHCS) - Evaluation of Efficacy, Safety, Plasma Levels and Evolution of Resistance
Brief Title: Raltegravir in the Swiss HIV Cohort Study
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: Swiss HIV Cohort Study (Network); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: SHCS Project No 564
Record Dates: First submitted 2009-05-18; First posted 2009-05-20 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: HIV Infection
Keywords: HIV; antiretroviral treatment; Swiss HIV Cohort Study; drug resistance; integrase inhibitor; Treatment
MeSH Terms: conditions — HIV Infections | interventions — Raltegravir Potassium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Within the framework of the Swiss HIV Cohort Study samples are taken of all patients regularly every 6 months. Plasma and frozen cells (www.shcs.ch)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Salvage group: In this group patients are enrolled that have failed previous antiretroviral drug regimens and qualify for Raltegravir treatment according to the approved indication of this drug in Switzerland.
  Interventions: Drug: Raltegravir
- Switch group: In this group, patients are enrolled which have to switch to Raltegravir due to drug toxicity or adverse events caused by other antiretroviral drugs.
  Interventions: Drug: Raltegravir

INTERVENTIONS:
Drug: Raltegravir — Raltegravir standard dosage of 400mg tablets every 12 hours together with an optimized backbone antiretroviral drug regimen
  Other Names: Isentress

SUMMARY:
Since June 2007, raltegravir has been available in Switzerland within a named patient program for patients who have virologic failure, triple class experience and resistance, and no other treatment options. This proposal has been designed to evaluate efficacy and safety data among patients who receive raltegravir within the routine clinical practice in Switzerland and who participate in the Swiss HIV Cohort Study. This is a combined retrospective analysis of patients who already received raltegravir and a prospective part of patients who enter the named patient program and will be followed up in a standardized way. In the prospective part, patients will also be able to receive raltegravir in case of intolerance to their current medication with virologic suppression.

The analysis will primarily use descriptive statistics. In addition, we will assess the duration of virologic response and focus on predictors of HIV RNA suppression during a follow-up of at least 6 months. In the prospective part, we will assess trough plasma levels of raltegravir and other antiretrovirals. In patients who will develop virologic failure, genotypic and phenotypic resistance to raltegravir (and other antiretrovirals) will be performed to characterize the evolution of resistance during the raltegravir-containing regimen.

ELIGIBILITY:
Inclusion Criteria:

* all patients treated with Raltegravir within the Swiss HIV Cohort Study

Exclusion Criteria:

* drop out of the Swiss HIV Cohort study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Swiss HIV Cohort study is a nationwide observational cohort existing for more than 20 years and is representative of the HIV-infected population in Switzerland (approx. 50% of HIV-infected patients in Switzerland, participate in this study). All patients must sign an informed consent to participate in this study.
  The study population enrolled in the current "Raltegravir in the SHCS" study, is a subgroup of patients, that has to go on Raltegravir within the Swiss HIV Cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2008-04; Primary Completion 2010-04 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
HIV RNA < 50 copies/ml | after 6 and 12 months

SECONDARY OUTCOMES:
durability of HIV RNA suppression | time to virological failure
predictors of HIV RNA suppression (viral load and CD4 at baseline, resistance at baseline for those with detectable HIV RNA, number of active drugs within the salvage regimen | baseline
time course of CD4 lymphocytes | baseline until study end
severe drug-related adverse events | during study period
drug levels of raltegravir and other antiretroviral drugs | during first year of Ral treatment
evolution of resistance in patients with virologic failure while on raltegravir | time to failure

CONTACTS AND LOCATIONS:
Overall Officials: Huldrych F Günthard, MD, Principal Investigator — University of Zurich, University Hospital of Zurich, Switzerland
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

REFERENCES:
- See also: Describes the Swiss HIV Cohort Study — http://www.shcs.ch